CLINICAL TRIAL: NCT04263155
Title: Implementation and Evaluation of the Peer-Delivered Body Project for Young Women in High School
Brief Title: The Peer-Delivered Body Project for Young Women in High School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Sona Dimidjian, Principal Investigator, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-0007-01
Record Dates: First submitted 2020-01-29; First posted 2020-02-10 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Eating Disorders in Adolescence
Keywords: Eating disorder prevention; Body Project; Female; Adolescence; Peer delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: The Body Project for high school young women (Experimental): The 4-hour Body Project workshop delivered by trained peer leaders
  Interventions: Behavioral: The Body Project
- Control (No Intervention): The business-as-usual comparison group does not participate in the Body Project but may engage in any other programs or services they normally would

INTERVENTIONS:
Behavioral: The Body Project — The Body Project is a 4-hour dissonance-based program designed to address body image concerns and prevent eating disorders. The curriculum consists of written, verbal, and behavioral exercises that provide participants with the opportunity to voluntarily and publicly critique the appearance ideal.
  Arms: Experimental: The Body Project for high school young women

SUMMARY:
This study will evaluate the impact of the Body Project (a dissonance-based program designed to address body image concerns and prevent eating disorders) on key eating disorder risk factors and relevant social and self-constructs at three time-points (pre, post, and one-year follow-up). Young women will be recruited from two high schools and will be randomized to receive the Body Project or to the control group. The Body Project will be facilitated by college-aged women.

DETAILED DESCRIPTION:
Preventive models that can avert the onset of eating disorders and innovative delivery methods that increase engagement with care offer a promising approach to improving the mental health and wellness of young women. This study aims to implement and evaluate the Body Project, a 4-hour dissonance-based program designed to address body image concerns and prevent eating disorders with high school young women using a peer delivery model. This study will evaluate the impact of the Body Project on key eating disorder risk factors and relevant social and self-constructs at three time-points (pre, post, and one-year follow-up). Young women will be recruited from two high schools and will be randomized to receive the Body Project program or to the control group. The Body Project will be facilitated by college-aged young women who have been trained to deliver the Body Project.

ELIGIBILITY:
Inclusion Criteria:

- Female high school student

Exclusion Criteria:

- Previous participation in the Body Project program

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 74 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Thin-Ideal Internalization Scale | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of endorsement of the thin ideal (scale 1-5 with higher scores indicating higher levels of thin ideal internalization)
Change in Satisfaction and Dissatisfaction with Body Parts Scale | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of body dissatisfaction (scale 1-5 with higher scores indicating higher levels of dissatisfaction)
Change in Dutch Restrained Eating Scale | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of dietary restraint (scale 1-5 with higher scores indicating higher levels of eating restraint)
Change in Positive Affect and Negative Affect Scale-Revised | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of negative affect (scale 1-5 with higher scores indicating higher levels of negative affect)

SECONDARY OUTCOMES:
Change in Objectified Body Consciousness Scale - Body Surveillance Subscale | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of body monitoring and surveillance (scale 1-7 with higher scores indicating higher levels of body surveillance)
Change in UCLA Loneliness Scale | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of loneliness (scale 1-4 with higher scores indicating higher levels of loneliness)
Change in Inventory of Peer Influence on Eating Concerns | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of peer influence on eating and body concerns (scale 1-5 with higher scores indicating higher levels of peer influence)
Change in Patient Health Questionnaire (PHQ-9) | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure for depressive symptom severity(scale 0-3 with higher scores indicating higher levels of depression)
Change in Generalized Anxiety Disorder (GAD-7) | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure for symptoms of generalized anxiety (scale 0-3 with higher scores indicating higher levels of anxiety)
Change in General Self-Efficacy Scale | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of self-efficacy (scale 1-4 with higher scores indicating higher levels of self-efficacy)
Change in Self-Compassion Scale | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of self-compassion (scale 1-5 with higher scores indicating higher levels of self-compassion)
Change in Rosenberg Self-Esteem Scale | Baseline, Post-intervention (4 weeks after baseline), 1 year post-intervention follow-up
  Self-report measure of global self-worth (scale 1-4 with higher scores indicating higher levels of self-esteem)
Sense of Belonging (Body Project group only) | Baseline
  Self-report measure of anticipated belonging with group (scale 1-7 with higher scores indicating higher levels of anticipated belonging)
Sense of Belonging Follow-Up (Body Project group only) | Post-intervention (4 weeks after baseline)
  Self-report measure of belonging with group (scale 1-7 with higher scores indicating higher levels of experienced belonging)
Working Alliance Inventory (Body Project group only) | Post-intervention (4 weeks after baseline)
  Self-report measure of therapeutic alliance with peer leaders (scale 1-5 with higher scores indicating higher levels of working alliance)
Program Satisfaction (Body Project group only) | Post-intervention (4 weeks after baseline)
  Self-reported ratings of satisfaction with program and peer leaders (scale 1-4 with higher scores indicating higher levels of program satisfaction)
Fidelity and Competence (Body Project group only) | From the first Body Project session to the final (fourth) Body Project session, 4 weeks on average
  Observer-rated assessments of peer leader fidelity and competence (scale 1-10 with higher scores indicating higher levels of facilitator fidelity and competence)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanderkruik R, Gist D, Dimidjian S. Preventing eating disorders in young women: An RCT and mixed-methods evaluation of the peer-delivered Body Project. J Consult Clin Psychol. 2020 Dec;88(12):1105-1118. doi: 10.1037/ccp0000609. PMID 33370134